CLINICAL TRIAL: NCT01792167
Title: Multi-site Evaluation of Second Step: Student Success Through Prevention (Second Step - SSTP) in Preventing Bullying and Sexual Violence
Brief Title: Multi-Site Evaluation of Second Step
Acronym: SSTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dorothy Espelage, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01CE001677 (NIH); UIUC 10147 (Other: Institutional Review Board)
Record Dates: First submitted 2012-03-07; First posted 2013-02-15 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Second Step (Experimental): Second Step Curriculum
  Interventions: Behavioral: Second Step Curriculum
- Stories of Us (No Intervention): Stories of Us was provided to schools

INTERVENTIONS:
Behavioral: Second Step Curriculum — social emotional learning program for 6th-8th graders. 15 50 minutes lessons in 6th grade, 13 50 minute lessons in 7th and 8th grade. covers empathy, perspective taking, anger management, impulse control, problem-solving, alcohol and drug prevention, sexual harassment, prejudice, bully prevention, bystander intervention
  Arms: Second Step

SUMMARY:
This study is a large-scale, randomized longitudinal evaluation of Second Step: Student Success Through Prevention (Second Step - SSTP), a middle school intervention (Committee for Children, 2008), which targets the shared underlying risk and protective factors for bullying, sexual harassment, and dating aggression. This program is unique in its emphasis on the role of peer group norms, attitudes, and behavior in the initiation and maintenance of bullying and other forms of violence. Because of this, this investigation will involve a direct test via social network analysis the extent to which peer norms or shifts in peer attitudes are impacted by the intervention. Bullying is conceptualized as including verbal, physical, relational, and cyber-aggression. Sexual violence is conceptualized as including sexual harassment, sexual coercion in dating relationships, and homophobic teasing. Thirty-six schools were drawn from four school districts in Illinois and one large district in Wichita, Kansas and randomly assigned to Second Step - SSTP or a control condition. Second Step -SSTP program draws from the risk/protective factors model and social-cognitive theories of aggression. Lessons focus on the outcomes of bullying, relational aggression, sexual harassment, dating relationships, and substance use. Risk factors targeted include inappropriate classroom behavior, favorable attitudes toward aggression and substance abuse, deviant peer affiliation, peer rejection, and impulsiveness are targeted as risk factors. Targeted protective factors include empathy, problem-solving skills, school connectedness, assertiveness and adoption of conventional norms. The P3R: Stories of Us - Bullying program, composed of a series of film-based education will be used in the control schools. All 6th graders at each school will be recruited and followed for the three year study period. Students and teachers will complete self-report and nomination tasks. Growth curve analysis via hierarchical linear modeling (HLM; Bryk & Raudenbush, 1992) will be utilized to assess change in the major dependent variables (bullying, sexual harassment perpetration, dating aggression), structural equation modeling will test for mediators across the study period, and social network analysis will be instrumental in identifying peer norms and attitudes.

DETAILED DESCRIPTION:
Seven outcome measures were evaluated including bullying perpetration, peer victimization, physical fighting, homophobic name calling (victimization and perpetration), and sexual violence (victimization and perpetration). Given that students in the intervention received only one-year (15 lessons; 50 minutes/week) of the developmentally-sequenced three-year curriculum, it was hypothesized that the strongest intervention effect would be seen for overt physical aggression, followed by more subtle effects for bullying and peer victimization outcomes. Because students were not introduced to concepts of prejudice, bias, and sexual violence (referred to sexual harassment) until the 7th and 8th grade curriculum, it was hypothesized that no significant intervention effects would emerge for these constructs at this point in time.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at one of our participating schools

Exclusion Criteria:

* None

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4089 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
aggression perpetration | pre (fall 2010), three posts (spring 2011, 2012, 2013)
  Using University of Illinois Fight Scale (Espelage & Holt, 2001)

SECONDARY OUTCOMES:
sexual violence | pre (fall 2010), 3 posts (spring 2011, 2012, 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy L Espelage, Ph.D., Principal Investigator — University of Illinois, Urbana-Champaign
Locations (1):
- University of Illinois, Champaign, Dept of Educational Psychology, Champaign, Illinois, United States